CLINICAL TRIAL: NCT03123666
Title: Randomized Controlled Trial of Recombinant Human Granulocye Monocyte - Colony Stimulating Factor (GM CSF) for Prevention of Pneumonia in Patients With Cirrhosis
Brief Title: Recombinant Human Granulocyte Monocyte - Colony Stimulating Factor (GM CSF) for Prevention of Pneumonia in Patients With Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-09
Record Dates: First submitted 2017-04-19; First posted 2017-04-21 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2019-12

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Granulocyte/macrophage colony-stimulating factor (GM-CSF) (Experimental): GM CSF (Sargamostatim-250mcg/M2) over 4 hour and inhalation of same dose by micronebulizer OR Placebo for 7 days. Both the groups will receive standard medical care
  Interventions: Drug: GMCSF
- Placebo (Placebo Comparator): Placebo will be given identical to the interventional
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GMCSF — GM CSF (Sargamostatim-250mcg/M2) over 4 hour and inhalation of same dose by micronebulizer
  Arms: Granulocyte/macrophage colony-stimulating factor (GM-CSF)
Other: Placebo — Placebo identical to GMCSF will be given
  Arms: Placebo

SUMMARY:
Informed consent obtained from the patient or the patient's legal surrogate. The window for randomization and initiation of study drug infusion is 2 days from day of Admission. All further time points are relative to the day of randomization. Patients will be randomized (1:1) to receive either recombinant human GM-CSF or placebo. Using randomized block design of 10 each generated by computer and provided in sequential, sealed, opaque envelopes. Subjects will be stratified based on Child status. Patients who fulfil the inclusion criteria will receive either slow IV infusion of GM CSF (Sargamostatim-250mcg/M2) over 4 hour and inhalation of same dose by micronebulizer for 7 days OR Placebo(saline infusion and saline nebulization). Standard medical care will be given in both limbs.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cirrhosis admitted to ICU-HDU without pneumonia at admission
* 18-70 years of Age
* Child B/ C

Exclusion Criteria:

* Patient having pneumonia
* If there is evidence of preexisting chronic respiratory failure
* If the patients is neutropenic (absolute neutrophil count <1000 cells/mm3
* If there was a history of hematological malignancy or bone marrow transplantation
* Person having HCC
* Acute liver Failure
* Pregnancy
* HIV

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2020-10-19 (Estimated); Study Completion 2020-10-19 (Estimated)

PRIMARY OUTCOMES:
Survival in both groups | 1 year

SECONDARY OUTCOMES:
Development of extra pulmonary organ failure during the course of study. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No